CLINICAL TRIAL: NCT07390344
Title: VIATORR® TIPS Study Evaluating 6-10mm Diameters (VIATIPS)
Acronym: VIATIPS
Status: Not yet recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: VTR 25-07
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ascites; Variceal Bleeding; Portal Hypertension Related to Cirrhosis
Keywords: portal hypertension; TIPS; cirrhosis; decompensated; Transjugular Intrahepatic Portosystemic Shunt
MeSH Terms: conditions — Ascites; Hypertension, Portal; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects treated for portal hypertension with the Registry device: The study population consists of patients treated with the GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion 6-10mm for portal hypertension and its complications including but not limited to variceal bleeding and/or ascites.
  Interventions: Device: GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion (6-10mm)

INTERVENTIONS:
Device: GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion (6-10mm) — The GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion (6-10mm) was developed and approved for the treatment of portal hypertension and its complications such as bleeding from enlarged or swollen veins (variceal bleeding) and abnormal build-up of fluid in the abdomen that does not respond to therapy (ascites which recurs despite conventional treatment).
  The Registry Device is a small tube (stent) that creates a pathway for blood flow. It consists of a metal frame (nitinol), covered with a thin, flexible material called expandable polytetrafluoroethylene (ePTFE).

SUMMARY:
This Registry will look at patients being treated with a transjugular intrahepatic portosystemic shunt (TIPS) procedure for portal hypertension. The purpose of this Registry is to collect data on the safety and performance of the GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion (6-10mm) for 2 years in real world setting.

Additionally, data will be collected on the safety and performance of the GORE TIPS Set when utilized.

DETAILED DESCRIPTION:
The GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion (6-10mm) was developed and approved for the treatment of portal hypertension and its complications such as bleeding from enlarged or swollen veins (variceal bleeding) and abnormal build-up of fluid in the abdomen that does not respond to therapy (ascites which recurs despite conventional treatment).

Subjects will receive the Registry Device as part of standard treatment for their condition. This means within this Registry, the information collected reflects the use of the Registry Device in typical, everyday medical practice by physicians, often referred to as "real world" data.

Patient total sample size will target a total approximately 152 patients treated with GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion (6-10mm).

Subjects who meet all criteria may be enrolled in the Registry.

The first visit after the procedure will be performed at the day of discharge or within 7 days after the procedure, whatever comes first. Subjects will have follow-up visits at 1 month, 3 months, 6 months, 12 months, and 24 months after their procedure so their health and the performance of the Registry Device can be monitored.

During follow-up visits, the doctor will perform a physical exam, review medications, and perform a condition status assessment. Imaging will not be collected as part of the Registry but may be ordered by the doctor for safety follow-up purposes as imaging is often collected as part of standard medical care.

Subjects will be asked to complete Quality of Life questionnaires at each follow-up visit to collect information on their well-being and daily life.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is eligible for treatment with the GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion 6-10mm for de novo TIPS creation.
2. The subject has cirrhotic portal hypertension.
3. The subject is ≥18 years of age.
4. The subject is capable of complying with protocol requirements, including follow up.
5. The subject or legal representative signed the informed consent form (ICF).

Exclusion Criteria:

1. The subject has any portal vein thrombosis, including both occlusive and non-occlusive thrombosis.
2. The subject has received a liver transplantation. Patients on the transplant list are still eligible.
3. The subject has a life expectancy of less than 6 months.
4. The subject has extrahepatic or hepatic malignancy or a history of previous malignancy, unless treated curatively ≥5 years prior to enrollment. Subjects with non-melanoma skin cancer and/or carcinoma in situ of the cervix remain eligible.
5. The subject has inadequate functional hepatic reserve with a Model for End-Stage Liver Disease (MELD) Score of > 25 or Child Pugh Score of > 14.
6. The subject is enrolled in another investigational study, unless agreed in advance in writing by the Sponsor.
7. The subject is pregnant at the time of informed consent signature.
8. The subject has any other condition which in the judgement of the investigator would preclude adequate Study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects treated with the GORE® VIATORR® TIPS Endoprosthesis with Controlled Expansion 6-10mm for portal hypertension and its complications including, but not limited to, variceal bleeding and/or ascites.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Subjects achieving primary patency through 2 years | Shunt primary patency will be analyzed at 1, 3, 6, 12 and 24 months.
  Freedom from shunt occlusion on imaging or from reintervention due to shunt dysfunction (occlusion or thrombosis on imaging or significant stenosis confirmed by venography).

SECONDARY OUTCOMES:
Proportion of Subject procedures that are a technical success | Day 0
  Successful delivery and deployment of the device to create an intrahepatic shunt connection between the portal and hepatic circulations.
Reduction in portosystemic gradient (PSG) | Day 0
  Difference between the pre-TIPS gradient (prior to TIPS device deployment) and the post-TIPS gradient (at completion of procedure).
Proportion of Subjects with variceal rebleeding through 2 years | Variceal rebleeding will be analyzed at 1, 3, 6, 12 and 24 months.
  Variceal rebleeding is defined as any endoscopically proven variceal bleeding event that occurs post procedure. The inability to control acute bleeding after device implant at time of procedure will count as a rebleeding event on day 0.
Rate of large volume paracentesis (LVP) through 2 years per subject-month | LVP frequency will be analyzed at 1, 3, 6, 12, and 24 months.
  Any reported episode of large volume (≥ 5 L) paracentesis following the TIPS procedure.
Change in Quality of Life from baseline | Baseline and 1, 3, 6, 12, and 24 months
  Change in Quality of Life as measured by the European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) and Chronic Liver Disease Questionnaire (CLDQ).